CLINICAL TRIAL: NCT03519334
Title: PArticipation To Healthy Workplaces And Inclusive Strategies in the Work Sector
Brief Title: PATHWAYS in Europe
Acronym: PATHWAYS
Status: Completed | Type: Observational
Sponsor: Maria Cabello (Other)
Collaborators: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); Ludwig-Maximilians - University of Munich (Other); Fundació Sant Joan de Déu (Other); University Rehabilitation Institute, Republic of Slovenia (Other); University of Thessaly (Other); KABEG Management (Other); Jagiellonian University (Other); Charles University, Czech Republic (Other); Oslo Metropolitan University (Other); European Association of Service providers for Persons with Disabilities (Unknown)
Responsible Party: Sponsor-Investigator, Maria Cabello, PhD, Universidad Autonoma de Madrid
Organization: Universidad Autonoma de Madrid (Other)
Other Study IDs: PATHWAYS2020; HP-PJ-2014-663474 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2017-11-08; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2017-11

CONDITIONS: Employment
Keywords: Employment; Return to work; Career Mobility; Employment supported; Workplace; Chronic disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic health condition group/study: People with any of the following chronic health conditions: Diabetes, Chronic obstructive Pulmonary Disease, Major Depression, Dysthymia, Migraine, Back & Neck Pain, Cancer, Ischemic Heart Disease
- Expert consultation group/study: Relevant contacts from advocacy organizations operating at European level for the professional integration of people with chronic health conditions.

SUMMARY:
PATHWAYS is a 3-year project that directly contributes to the 2014 Work Programme by focusing on action 2.1.1.3 regarding the development of innovative approaches to promote the professional integration and reintegration of people with chronic diseases and improve their employability. The main aim of PATHWAYS is to provide evidence-based recommendations for the effective professional integration of people with chronic health conditions in Europe

DETAILED DESCRIPTION:
Introduction: One out four people experience any long-lasting health problem in Europe. Individuals with chronic diseases often experience work-related problems, leading to negative consequences at individual and societal level. The rising prevalence of chronic diseases as well as the current economic recession made this issue even more problematic, requiring action in terms of innovative strategies to improve the participation of these persons in the labor market.

The PATHWAYS objectives are:

1. To identify integration and re-integration strategies that are available in Europe and beyond and to determine their effectiveness (systematic literature review)
2. To assess the specific employment related needs of persons with chronic diseases and mental disorders (e-survey including people with chronic health conditions)
3. To develop guidelines supporting the implementation of effective professional integration and reintegration strategies. (expert consultation survey)

Methods:

PATHWAYS is a multi-informant approach study. Information will be gathered from different sources:

1. Systematic literature review,
2. An expert consultation study (Including NGOs, patient's organizations and advocacy organizations operating at European Level). Experts will be searched by Internet. Questionnaire will be completed by e-mail
3. an e-Survey including people with chronic health conditions. The Clinical Record Form (CRF) will be online (Google forms). Participation will be free. Any people who meet the inclusion criteria can log in and complete it. The dissemination of the CRF will be done via relevant patient's associations. The CRF will be also published in the patient association's websites, if possible

Hypothesis:

* Literature will focus on the negative points of experiencing chronic health problems in the workplace rather than analysing the professional needs of people with these health conditions
* There will be a set of professional needs that will be shared across different chronic health condition groups and that can be targeted in common preventive strategies
* There will be a considerable gap between the existing employment strategies (i.e. services, systems and policies) and the real employment needs of people with chronic health conditions

ELIGIBILITY:
As PATHWAYS include different studies and methodologies, different inclusion and exclusion criteria are defined for each study

People with Chronic health condition study:

Inclusion Criteria:

* People with self-reported diagnosis of chronic health conditions (i.e Diabetes, Chronic obstructive Pulmonary Disease, Major Depression, Dysthymia, Migraine, Back & Neck Pain, Cancer, Ischemic Heart Disease)
* Participants living in European Union (EU-28)
* Working age: 18-65 years

Exclusion Criteria:

* Younger than 18 years
* No residents in European Union (EU-28)

Expert consultation study:

Inclusion Criteria:

* People working in Advocacy organizations. These organizations should meet all the following criteria: i) their main activities should be addressed at (re)integrating people with chronic health conditions into the workforce ii) they should operate at European level, and iii) they should have at least 3 years of experience in the field.
* Working age: 18-65 years

Exclusion Criteria:

* Advocacy organizations not operating at European Union Level

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic health conditions will be defined by people with self reported diagnosis of any of the following health conditions: Diabetes, Chronic obstructive Pulmonary Disease, Major Depression, Dysthymia, Migraine, Back & Neck Pain, Cancer, Ischemic Heart Disease (According to International Classification of Diseases 10th version (ICD-10)
  Experts will be people working in advocacy organizations. For example, NGOs and patient's associations. These associations shuld be aimed ar enhancing professional integration of people with chronic health conditions
Sampling Method: Non-Probability Sample
Enrollment: 686 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Employment needs | One time point assessment. Period of data collection: An average of 3 years (2016-2018)
  Any environmental or personal factor that impact on the professional integration of people with chronic health conditions. This definition has been conceptualized according to the International Classification of Disability and Health's framework (World Health Organization, 2001). This outcome will be collected in the e-survey study (including people with chronic health conditions)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Mateos, MD, PhD, Principal Investigator — Universidad Autonoma de Madrid
Locations (10):
- KABEG Gailtal-Klinik, Hermagor, Austria
- Charles University Czech Republic, Prague, Czechia
- Ludwig Maximilian University, Munich, Germany
- University of Thessaly, Thessaloniki, Greece
- Foundation IRCCS Neurological Institute Carlo Besta, Milan, Italy
- Oslo and Akershus University College of Applied Sciences, Oslo, Norway
- Jagiellonian University Medical College, Krakow, Poland
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia
- Spain (2):
  - Fundació Sant Joan de Déu, Sant Boi de Llobregat, Barcelona
  - Universidad Autonoma de Madrid, Madrid

IPD SHARING:
Plan to Share IPD: Undecided
A sharing plan description has to be still agreed between different Principal Investigators

REFERENCES:
- See also: PATHWAYS website — http://path-ways.eu/